## **Exhibit A: Study Services and Compensation**

| Title | Complications and 1-Year Outcomes following hiatal hernia repair with MIROMESH a novel, highly vascular, porcine derived, biologic matrix |
|---|---|
| Miromatrix<br>Product | MIROMESH® Biologic Matrix |
| Sponsor | Miromatrix Medical Inc<br>10399 W. 70 <sup>th</sup> Street<br>Eden Prairie, MN 55344 |
| Protocol Number | 2017001 Version 2 |
| Sponsor Contact | M. Mason Macenski, Ph.D.<br>952.942-6000 X112<br>612.378-2612 |
| Principal<br>Investigator | G. Kevin Gillian, MD |
| Study Center | Virginia Heartburn and Hernia Institute<br>8988 Lorton Station Blvd<br>Suite 202<br>Lorton, VA 22079 |
| Planned Sample<br>Size | 70 consecutive subjects at least 1-year post-index procedure |
| Study Population | Consecutive cohort of patients who have undergone a hiatal hernia repair between 1 Jul 2015 and 1 June 2016 • A <i>minimum</i> of three attempts to reach each subject in the cohort shall be made |
| Study Objectives | Primary Objective |
| | Characterize the procedural and early post-operative safety profile of MIROMESH when used as reinforcement in hiatal hernia repair. |
| | Secondary Objectives |
| | Identify a consecutive cohort who may be tracked long term to identify survival of repair. Identify a consecutive cohort who may be tracked long term to characterize mid- and long-term clinical outcomes. |
| | Identify a consecutive cohort who may be tracked long term to further characterize the safety profile over time. |
| Study Design | This will be a retrospective chart review to identify the appropriate cohort with a prospective follow-up survey to acquire safety and outcome information. |
| Study Assessments and Time Points | Preoperative – Chart Review A retrospective chart review of appropriate subjects. Data to be acquired will be: Gender Date of birth Weight BMI |

| | Specific diagnosis |
|---|---|
| | DeMeester Score |
| | • 24 hour <i>pH</i> test (% acid exposure in 24 hours) |
| | GERD-HRQL Score |
| | Peri-operative Preoperative — Chart Review |
| | Date of surgery |
| | Number of stitches used to close wound |
| | Paraesophageal hernia type |
| | Mesh shape |
| | Mesh size used |
| | Attachment technique |
| | Length of stay |
| | Complications |
| | Post-Operative (With-in 1 month of surgery) Preoperative — Chart Review |
| | Complications (Mesh related) |
| | Complications (Mesh related) Complications (procedure related) |
| | Prolonged dysphagia (Y/N) |
| | Stenosis (Y/N) |
| | Dilations (Y/N) |
| | EGD/UGL documented hernia recurrence |
| | GERD-HRQL Score |
| | Minimum 1-year Follow-Up Telephone Interview |
| | Have you had a revision surgery? |
| | GERD-HRQL Score |
| | <ul> <li>How satisfied are you with the procedure?</li> </ul> |
| | How likely are you to recommend this procedure to a loved one? |
| Timeline | Data collection will be complete 3-months after approval and funding |
| Assessment Tools | Patient Charts |
| | DeMeester Score |
| | 24 hour <i>pH</i> test (% acid exposure in 24 hours) |
| | GERD-HRQL Score |
| Project Budget | \$15,000 and IRB fees as invoiced (or directly paid) |
| . reject Budget | 25% upon full execution of agreement |
| | 25% Upon receipt of spreadsheet showing 50% (35 subjects) |
| | completion |
| | 25% upon receipt of spreadsheet with all subject data (70 subjects) |
| | 25% upon receipt of study report – narrative style |
| Privacy | Principle Investigator and Sponsor will enter into a Limited-Data Set Data Use |
| Considerations | Agreement consistent with 45 CFR 164.514. Data listed above will be |
| | transferred and no protected health information not specifically covered by the |
| | data use agreement will be delivered to the sponsor. |
| Informed Consent | All subjects will be required to give verbal consent, via the telephone interview, |
| | for participation in this study. Subjects will be informed that they were chosen |
| | · |

| | based on the procedure and mesh they received. They will be informed that historical data regarding their pathology and procedure will be gathered and that they will be asked several questions about their current health. They will be informed that, except for, information used to determine age and date of surgery, no protected health information will be used. Subjects that elect to participate will be informed that they will receive a copy of the verbal informed consent. Investigator will mail a copy of the consent script to all subjects who elect to participate in this study. |
|---|---|
| Ethical<br>Considerations | This Study Proposal Summary will be reviewed by an accredited institutional review board and will not be initiated until written approval has been received. |
| Statistical Analysis | Descriptive statistics including but not limited to mean, standard deviation, frequency and percentages will be used to describe demographics, medical history, and characterize baseline variable as appropriate. Inferential statistics will be used to describe changes in variable over time. |
| Deliverable(s) | Excel spreadsheet with all data as outlined above Narrative study report outlining results and drawing conclusions. |